CLINICAL TRIAL: NCT05358990
Title: Knowledge Mobilization Activities to Support Decision-making by Youth, Parents and Adults Using a Systematic and Living Map of Evidence and Recommendations on Coronavirus Disease (COVID-19)
Brief Title: Knowledge Mobilization Activities to Support Decision-Making by Youth, Parents and Adults: Study Protocol
Acronym: eCOVID-PLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Western University (Other); The Hospital for Sick Children (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Holger Schunemann, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 3856
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: electronic Coronavirus Disease Recommendation Map (eCOVID RecMap); Plain Language Recommendation; Standard Language Versions; Public Engagement; Knowledge Mobilization
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plain Language Recommendation (PLR) (Experimental): New easy to read COVID-19 recommendations available on the COVID19 Living Map of Recommendations and Gateway to Contextualization (RecMap).
  Interventions: Other: Plain Language Recommendation (PLR)
- Standard Language Version (SLV) (Active Comparator): Original recommendation as initially published by the guideline organization.
  Interventions: Other: Standard Language Version (SLV)

INTERVENTIONS:
Other: Plain Language Recommendation (PLR) — New easy to read COVID-19 recommendations available on the COVID19 Living Map of Recommendations and Gateway to Contextualization (RecMap).
  Arms: Plain Language Recommendation (PLR)
Other: Standard Language Version (SLV) — Original recommendation as initially published by the guideline organization.
  Arms: Standard Language Version (SLV)

SUMMARY:
Coronavirus Disease (COVID-19) recommendations are usually developed for healthcare professionals (for example Doctors, health organizations, etc.). It is important to make sure that these recommendations can be used and understood by everyone. This study aims to make COVID-19 recommendations more accessible and understandable for parents and caregivers, adults, and youth.

DETAILED DESCRIPTION:
This is a two-arm superiority randomized controlled trial. The primary objective is to compare the understanding of key guideline information between the Plain Language Recommendation (PLR) (intervention) and the Standard Language Version (SLV- original recommendation as available in the published guideline) (comparison). Secondary outcomes include accessibility and usability of the information, satisfaction with the presentation, intended behavior to follow the information in the recommendation, and preference toward one of the two presentations. Recruitment will be global for the three populations (youth, parents, and adults), using three different online links. Data will be collected using a survey with 1:1 randomization to the intervention and subsequent demographic questions. Superiority will be declared if a minimal difference of 10% in understanding is achieved between the two groups (an average difference of 1 correct answer).

ELIGIBILITY:
Inclusion Criteria:

* For youth population: be between the ages of 15 to 24 years
* For parents population: be 18 years and above and making decisions with or for their children (parent, caregiver, the legal guardian of a child < 18 years)
* For adults: be 21 years of age or older
* Need to be able to complete the survey in English

Exclusion Criteria:

* Individuals not fitting any of the above age categories or language requirement

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 997 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Understanding with Multiple Choice Questions | Duration of survey (approximately 25 minutes) at baseline
  The primary outcome is understanding. Understanding is defined as the correct comprehension of key guideline content (year of publication, intent of the recommendation, direction of recommendation, etc.). This outcome will be measured with seven multiple-choice questions about key concepts in the recommendation with four to six response options for each question and only one correct answer (total minimum score of 0, maximum score of 7).

SECONDARY OUTCOMES:
Accessibility and Usability on a Seven-Point Likert Scale | Duration of survey (approximately 25 minutes) at baseline
  Accessibility and Usability is defined as the ability to find/access, and use the presented information. This outcome considers the three following domains: (1) how easy it was to find information, (2) how easy it was to understand the information (perception), and (3) whether the information was presented in a way that could be helpful for making an informed health decision. Participants will have to indicate the degree of agreement with six statements, measured using the original 7-point Likert scale (1 being strongly disagree, 4 being neutral, and 7 being strongly agree). The outcome 'overall accessibility of information' will be measured using the 7-point Likert-type scale.
Satisfaction on a Seven-Point Likert Scale | Duration of survey (approximately 25 minutes) at baseline
  Satisfaction is defined as participants' impression of the recommendation's presentation. This will be measured using questions related to participants' level of satisfaction with the different features of the format (e.g. feature of explaining the certainty of the evidence). Participants will have to indicate the degree of satisfaction with three questions measured using the original 7-point Likert-type scale (11 = very dissatisfied, 2 = dissatisfied, 3 = somewhat dissatisfied, 4 = neutral, 5 = somewhat satisfied, 6 = satisfied, 7 = very satisfied). Participants will also have to answer three open-ended questions to get their input on what they liked and disliked in the format.
Intended Behavior on a Seven-Point Likert Scale and Multiple Choice Questions | Duration of survey (approximately 25 minutes) at baseline
  Intended behavior is defined as participants' intention in adopting and following the shared recommendation. Participants will answer a question on whether they have already followed and implemented the recommendation in their jurisdiction and have them respond with yes, no, unsure, or not applicable. Subsequently, they will be asked how likely it is that they will follow and share the recommendation through two questions measured using a 7-point Likert-scale (1 = very unlikely, 2 = unlikely, 3 = somewhat unlikely, 4 = neutral, 5 = somewhat likely, 6 = likely, 7 = very likely.
Preference on a Seven-Point Likert-Scale | Duration of survey (approximately 25 minutes) at baseline
  Preference is defined as a greater liking of one format over the other (PLR or SLV). All participants will get to compare the optimized PLR and the SLV; after having completed the tasks in the group they were randomized to, participants will review the alternative format and indicate their preference for one of the two formats using a 7-point Likert-type scale (1 = strongly prefer SLV, 2 = prefer SLV, 3 = somewhat prefer SLV, 4 = same preference for SLV and PLR, 5 = somewhat prefer PLR, 6 = prefer PLR, 7 = strongly prefer PLR).

CONTACTS AND LOCATIONS:
Overall Officials: Holger J Schunemann, MD, PHD, Study Chair — McMaster University; Kevin Pottie, Principal Investigator — Western University; Martin Offringa, Principal Investigator — The Hospital for Sick Children Research Institute; Nancy Butcher, Principal Investigator — The Hospital for Sick Children Research Institute; Lisa Hartling, Principal Investigator — University of Alberta
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stallwood L, Sammy A, Prebeg M, Relihan J, Baba A, Charide R, Sayfi S, Elliott SA, Hartling L, Munan M, Richards DP, Mathew JL, Kredo T, Mbuagbaw L, Motilall A, Scott SD, Klugar M, Lotfi T, Stevens AL, Pottie K, Schunemann HJ, Butcher NJ, Offringa M; RecMap Members. Plain Language vs Standard Format for Youth Understanding of COVID-19 Recommendations: A Randomized Clinical Trial. JAMA Pediatr. 2023 Sep 1;177(9):956-965. doi: 10.1001/jamapediatrics.2023.2686. PMID 37548983
- [Derived] Elliott SA, Scott SD, Charide R, Patterson-Stallwood L, Sayfi S, Motilall A, Baba A, Lotfi T, Suvada J, Klugar M, Kredo T, Mathew JL, Richards DP, Butcher NJ, Offringa M, Pottie K, Schunemann HJ, Hartling L. A multimethods randomized trial found that plain language versions improved parents' understanding of health recommendations. J Clin Epidemiol. 2023 Sep;161:8-19. doi: 10.1016/j.jclinepi.2023.06.018. Epub 2023 Jul 6. PMID 37421995
- [Derived] Charide R, Stallwood L, Munan M, Sayfi S, Hartling L, Butcher NJ, Offringa M, Elliott S, Richards DP, Mathew JL, Akl EA, Kredo T, Mbuagbaw L, Motillal A, Baba A, Prebeg M, Relihan J, Scott SD, Suvada J, Falavigna M, Klugar M, Lotfi T, Stevens A, Pottie K, Schunemann HJ. Knowledge mobilization activities to support decision-making by youth, parents, and adults using a systematic and living map of evidence and recommendations on COVID-19: protocol for three randomized controlled trials and qualitative user-experience studies. Trials. 2023 Jan 14;24(1):27. doi: 10.1186/s13063-023-07067-9. PMID 36641457